CLINICAL TRIAL: NCT04275492
Title: Study on Bioequivalence of Pramipexole Dihydrochloride Sustained Release Tablets
Acronym: PLKS-BE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor terminated the clinical trial
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Hongguan biological pharmaceutical co. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ZYYY-PLKS-BE-2019-02
Record Dates: First submitted 2019-11-18; First posted 2020-02-19 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2019-11

CONDITIONS: Parkinson's Disease
Keywords: Pramipexole Dihydrochloride Sustained Release Tablets
MeSH Terms: conditions — Parkinson Disease | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting group (Experimental): Subjects were randomly assigned to one of two sequential groups (t-r group, r-t group) in a 1:1 ratio.In the first cycle, 15 subjects were given 1 tablet of test preparation (T) orally and 240mL warm water on an empty stomach, and the other 15 subjects were given 1 tablet of reference preparation (R, Siforl®) orally and 240mL warm water on an empty stomach.Cross-administration at 7±1 days.The authorized drug dispenser assigned the study drug to each phase of the study according to a randomized protocol.
  Interventions: Drug: Praxol hydrochloride sustained release tablet Specification: 0.375mg/ tablet (in pramipexole hydrochloride); Drug: Pramipexole hydrochloride sustained-release tablet (Siforl®) Specification: 0.26mg/ tablet (in pramipexole)
- Feeding group (Experimental): Subjects were randomly assigned to one of two sequential groups (t-r group, r-t group) in a 1:1 ratio.In the first cycle, 15 subjects took 1 tablet of the test preparation (T) orally and 240mL warm water about 30min after the high-fat meal, and another 15 subjects took 1 tablet of the reference preparation (R, Siforl®) orally and 240mL warm water about 30min after the high-fat meal.Cross-administration at 7±1 days.The authorized drug dispenser assigned the study drug to each phase of the study according to a randomized protocol.
  Interventions: Drug: Praxol hydrochloride sustained release tablet Specification: 0.375mg/ tablet (in pramipexole hydrochloride); Drug: Pramipexole hydrochloride sustained-release tablet (Siforl®) Specification: 0.26mg/ tablet (in pramipexole)

INTERVENTIONS:
Drug: Praxol hydrochloride sustained release tablet Specification: 0.375mg/ tablet (in pramipexole hydrochloride) — Praxol hydrochloride sustained release tablets, 0.375mg/ tablet, are manufactured by hongguanbio pharmaceutical co., LTD
Drug: Pramipexole hydrochloride sustained-release tablet (Siforl®) Specification: 0.26mg/ tablet (in pramipexole) — Siforl® is produced by Boehringer Ingelheim International Gmbh

SUMMARY:
The main purpose of In two kinds of fasting and postprandial Chinese healthy subjects with Boehringer represent Ingelheim company production of hydrochloric acid Pramipexole zyban (specification: 0.26 mg/piece, in Pramipexole, commodity name: Siforl ®) as the reference preparation, study a single oral dose of macro crown biological pharmaceutical co., LTD. Production of Pramipexole Dihydrochloride Sustained Release Tablets (specification:The pharmacokinetic parameters of the drug were calculated after the time course of the drug in vivo (0.375mg/ tablet, as measured by pramipexole hydrochloride), and the human relative bioavailability of the two preparations were compared to evaluate their bioequivalence.

A secondary purpose To evaluate the safety of fasting and postprandial oral test preparations and reference preparations.

DETAILED DESCRIPTION:
In this study, a single-center, randomized, open, two-cycle, self-crossover, single-dose administration design was used to evaluate the bioequivalence of the tested preparations and reference preparations given to Chinese healthy subjects with single-dose, fasting and post-meal administration of Pramipexole Dihydrochloride Sustained Release Tablets.

This study was divided into two parts: fasting administration and high-fat post-meal administration.The healthy subjects were randomly divided into two groups with the same number of patients in each group. The washing period was 7±1 days.

In this study, venous blood was collected at 18 time points (fasting and postprandial) within 1h (0h) before administration and at 1.0h, 2.0h, 3.0h, 4.0h, 5.0h, 6.0h, 7.0h, 8.0h, 9.0h, 10.0h, 11.0h, 12.0h, 16.0h, 36.0h, 48.0h, and 72.0h after administration.

A total of 60 healthy subjects were enrolled into the equivalence test, among which:

1. Study on human bioequivalence of drug administration on an empty stomach: 30 healthy subjects (male and female).
2. Human bioequivalence of high-fat post-meal administration: 30 healthy subjects (male and female).

ELIGIBILITY:
Inclusion Criteria:

* Subjects are fully aware of the purpose, nature, methods, and possible adverse effects of the test, volunteer as a subject, and sign the informed consent form before the start of any research program, and ensure that any program will be involved in the study;
* Male and female subjects aged 18-45 years (including 18 and 45 years)；
* Male body weight ≥50.0 kg, female body weight ≥45.0 kg;Body mass index [BMI= weight (kg)/ height (m)2] is within the range of 19.0~26.0 kg/m2 (including critical value)；
* According to the previous medical history, vital signs, comprehensive physical examination and required laboratory examination, the investigator determines that the patient is a healthy subject;
* Fully understand the purpose of the test, the nature of the test, the research procedures and possible adverse reactions, voluntarily participate in the test and sign the informed consent (the process of obtaining the informed consent conforms to the GCP regulations);
* The subject will be able to communicate well with the investigator, understand and comply with the requirements of this study, and be willing to be admitted to the phase I clinical research ward as required.

Exclusion Criteria:

* Have a history of allergy to this drug component or similar species;Had a history of allergy to two or more drugs, food, etc.;
* Have a history of dysphagia or any gastrointestinal diseases that affect drug absorption;
* Patients with any history of clinically serious diseases, including but not limited to diseases of digestive system, cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, neuropsychiatric system, blood system, immune system and metabolic abnormalities, which are clinically significant as judged by the investigator;
* Those who cannot tolerate venipuncture and have a history of acupuncture and blood sickness;
* Those who have received surgery (except appendicitis) within 3 months before screening, or who plan to have surgery during the study, and those who have received surgery that will affect drug absorption, distribution, metabolism and excretion;
* Screening those who had a history of drug abuse within the previous 6 months;
* Used drugs within 3 months before screening;
* Have participated in clinical trials of other drugs within 3 months before administration;
* Screening for blood donation within the first 3 months, including ingredient blood or massive blood loss (≥200mL), who received blood transfusion or used blood products;
* Have used any prescription drugs, non-prescription drugs, Chinese herbal medicine and vitamins within 2 weeks before administration;
* Those who smoked more than 5 cigarettes per day in the first 3 months or could not stop using any tobacco products during the trial;
* Those who drank more than 14 units of alcohol per week (1 unit of alcohol ≈360 mL beer or 45 mL spirits with a 40% alcohol content or 150 mL wine) in the first 3 months or who could not abstain from alcohol during the trial;
* People who drank excessive amounts of tea, coffee and/or caffeine-rich beverages (more than 8 cups, 1 cup =250 mL) every day for 3 months before screening;Or within 48 hours before the test, eat any food containing alcohol or rich in xanthine compounds (such as chocolate) and drink (such as tea, coffee, cola, etc.), grapefruit juice, etc；
* Lactose intolerant;
* Those who have special requirements on diet and cannot accept a uniform diet;
* The test of hepatitis b surface antigen, hepatitis c virus antibody, anti-human immunodeficiency virus antibody or anti-syphilis spirochete specific antibody has one or more clinical significance;
* Women who have positive pregnancy test results and are lactating, pregnant or planning to have a recent pregnancy;
* Those with positive alcohol test results or positive screening for drug abuse (morphine, methamphetamine, ketamine, dimethylene dioxymethamphetamine and tetrahydrocannabinic acid);
* Other subjects deemed unsuitable by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Cmax | [time range: 72 hours post-dose on Day 1,8]
  Maximum observed plasma concentration
Tmax | [time range: 72 hours post-dose on Day 1,8]
  Time to maximum plasma concentration
AUC（0-inf） | [time range: 72 hours post-dose on Day 1,8]
  Area under a time curve of plasma concentration from time 0 to infinity
AUC（0-72h） | [time range: 72 hours post-dose on Day 1,8]
  Area under the concentration-time curve 0 to 72 h after administration

CONTACTS AND LOCATIONS:
Overall Officials: Jian Liu, Master, Study Chair — The First Affiliated Hospital,ZheJiang Univercity
Locations (1):
- The First Affiliated Hospital,ZheJiang Univercity, Hanzhou, Zhejiang, China